CLINICAL TRIAL: NCT01319461
Title: Efficacy and Safety of Intraarticular Injections of Hyalgan in the Treatment of Osteoarthritis of the Knee: a Randomized, Masked Observed, Double Blind, Placebo Controlled, Multicenter Clinical Trial.
Brief Title: Efficacy and Safety of Intraarticular Injections of Hyalgan in the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Med Pharma Co., Ltd. (Industry)
Collaborators: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Eric Chang, Med Pharma Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UH-HYA-01-04
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Hyalgan
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sterile normal saline injection (Placebo Comparator)
  Interventions: Device: sterile normal saline
- Hyalgan injection (Experimental)
  Interventions: Device: Hyalgan

INTERVENTIONS:
Device: Hyalgan — Patients will receive intraarticular injection of 20mg /2ml /syringe Hyalgan® once a week for 5 consecutive weeks.
  Arms: Hyalgan injection
Device: sterile normal saline — Patients will receive intraarticular injection of sterile normal saline once a week for 5 consecutive weeks.
  Arms: sterile normal saline injection

SUMMARY:
Evaluate the efficacy and safety of Hyalgan, at a dose of 20mg/2ml administered as 5 intraarticular injections at weekly intervals, for the sustained relief of pain and amelioration of joint dysfunction in patients of OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female patients whose specific ages are > 50 years old, in general health. 2.Must be ambulatory (assistive devices allowed) 3.Patient was diagnosed as OA of knee joint by American College of Rheumatology (ACR) criteria ; [ ie,knee pain, and any one of the following:age>50 years,crepitus, or morning stiffness<30 minutes in duration ] 4.Radiographic confirmation of OA with Kellgren-Lawrence Ⅱ-Ⅲ score (mild to moderate)at the target joint (anterior-posterior views) with predominance in the tibia-femoral compartment 5.VAS score ≧40 mm for 50 foot of walking pain.

Exclusion Criteria:

* 1.Patients with severe degeneration of knee joint with marked joint narrowing, marked varus or valgus deformity of the knee greater than 12 o. 2.Patients with hepatic or renal failure, or other chronic severe diseases that can interfere with the outcome. 3.A known history of psychiatric diseases, significant neurological diseases, allergy or sensitivity to hyaluronic acid or avian protein. 4.Patients receive steroid intraarticular injection, anti-inflammatory agents less than two weeks. 5.Patients with joint disorders: inflammatory joint disease, specific arthropathy (chondrocalcinosis, joint effusion >30ml), severe axis deviations or instabilities, joint or skin infections, joint prostheses of the lower limbs, symptomatic hip. 6.Significant alcohol, drug or medication abuse as judged by the investigator. 7.Pregnancy determined by clinical evaluation or urine testing for nursing women and/or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm or Norplant). 8.Patients who have taken any other "investigational" drug within one month prior to the screening visit.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2001-05; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ching Tsai, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National taiwan university hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Huang TL, Chang CC, Lee CH, Chen SC, Lai CH, Tsai CL. Intra-articular injections of sodium hyaluronate (Hyalgan(R)) in osteoarthritis of the knee. a randomized, controlled, double-blind, multicenter trial in the Asian population. BMC Musculoskelet Disord. 2011 Oct 6;12:221. doi: 10.1186/1471-2474-12-221. PMID 21978211